CLINICAL TRIAL: NCT00500006
Title: A Phase I Dose Escalation of MK0457 in Combination With Dasatinib in Patients With Chronic Myelogenous Leukemia and Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: A Phase I Dose Escalation Combination Study in Patients With Chronic Myelogenous Leukemia (CML) and Philadelphia Chromosome-Positive (Ph+) Acute Lymphoblastic Leukemia (ALL)(0457-009)(TERMINATED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0457-009; 2007_509
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Myelogenous Leukemia; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tozasertib; Dasatinib

ARMS (2):
- A (Other): Arm A: Drug and comparator
  Interventions: Drug: MK0457; Drug: dasatinib
- B (Other): Arm B: Drug and comparator
  Interventions: Drug: MK0457; Drug: dasatinib

INTERVENTIONS:
Drug: MK0457 — Schedule A: 5-day continuous IV infusion every 28 days MK0457 (dose determined by height and weight). Starting dose = 20 mg/m2/hour titrating up to 33 mg/m2/hour.
  Schedule B: 6-hr IV infusion every 14 days MK0457 (dose determined by height and weight). Starting dose = 64 mg/m2/hour titrating up to 216 mg/m2/hour.
Drug: dasatinib — Oral dasatinib 70 mg b.i.d. tablets twice daily.
  Other Names: Sprycel®

SUMMARY:
This study will evaluate MK0457 in combination with Dasatinib in patients with Chronic Myelogenous Leukemia and Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia. Efficacy and Safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have chronic myelogenous leukemia (CML) or Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL)
* Patients must be at least 3 months from the start of dasatinib therapy and are currently receiving dasatinib therapy for CML or Ph+ ALL and be evaluable for hematologic response prior to entering the study
* Patient is able to be treated with a 70 mg bid dose of dasatinib without significant toxicity at the time of study entry
* Patients with active CNS disease are included and may be treated concurrently with intrathecal therapy as per institutional standards

Exclusion Criteria:

* Patient has had treatment with any anti-leukemia therapy (investigational or approved) other than dasatinib during the preceding 3 months. Pheresis or hydroxyurea treatment in the preceding 3 months will not exclude patients from eligibility
* Patient has unresolved more than or equal to grade 2 clinically significant toxicity attributed to dasatinib at the time of study entry
* Patient has known hypersensitivity to the components of study drug or its analogs
* Patient is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study
* Patient has symptomatic ascites, pericardial or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible
* Patient has had prior radiation therapy to more than 10% of the bone marrow; patients must have recovered for at least 3 weeks from the hematologic toxicity of prior radiotherapy
* Patient has a LVEF <40% by multigated radionucleotide angiography (MUGA) or echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, Safety, Tolerability | 28 Days

SECONDARY OUTCOMES:
Pharmacodynamics, Hematologic Response, Cytogenetic Response, Molecular Response, Response Durability | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Okabe S, Tauchi T, Ohyashiki K. Efficacy of MK-0457 and in combination with vorinostat against Philadelphia chromosome positive acute lymphoblastic leukemia cells. Ann Hematol. 2010 Nov;89(11):1081-7. doi: 10.1007/s00277-010-0998-x. Epub 2010 Jun 20. PMID 20563869